CLINICAL TRIAL: NCT05846165
Title: InveStigAting Bladder fiELd-cycLing imAging (ISABELLA)
Brief Title: InveStigAting Bladder fiELd-cycLing imAging
Acronym: ISABELLA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants identified. Funding ended
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2-115-22
Record Dates: First submitted 2023-03-29; First posted 2023-05-06 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; Bladder tumours; Field-Cycling Imaging
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bladder tumours (Experimental): Participants with muscle-invasive and non-muscle invasive bladder tumours of at least 3 cm in diameter will undergo one FCI scan.
  Interventions: Device: Field-Cycling Imaging (FCI)

INTERVENTIONS:
Device: Field-Cycling Imaging (FCI) — FCI scan

SUMMARY:
The goal of this pilot study is explore the parameters that can be obtained in bladder tumours by Field-Cycling Imaging (FCI) in patients with both muscle-invasive and non-muscle invasive tumours. The main question it aims to answer is if FCI can give more diagnostic information than conventional tests.

Participants will have one FCI scan and the results will be correlated with the results of CT urogram or CT scan.

DETAILED DESCRIPTION:
Patients with organ-confined muscle invasive bladder cancer are treated either by removal of their bladder at cystectomy or by organ-preserving treatment, generally following neoadjuvant chemotherapy. In some cases, the neoadjuvant chemotherapy can shrink the tumour so that it is clinically undetectable but there may still be tumour cells present microscopically. This presents a difficulty during planning of radiotherapy treatments, which could then miss the tumour and lead to tumour recurrence.

Field-Cycling Imaging (FCI) is an emerging imaging technology pioneered at the University of Aberdeen. FCI can image human tissues non-invasively over a wide range of magnetic field strengths, directly informing on multi-scale tissue structure from nanometres to micrometres. FCI has already shown significant potential for enhanced diagnosis in a range of diseases, and recent results show several potential biomarkers of cancer in breast, colon, and brain.

FCI has not been used in bladder cancer before. In this proof-of-concept study, we will recruit patients with both muscle-invasive and non-muscle invasive tumours to explore the parameters that can be obtained in bladder tumours by FCI. Results of the FCI scans will be correlated with the results of CT urogram or CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending for flexible cystoscopy found to have a tumour of at least 3 cm in diameter (muscle-invasive or non-muscle invasive)
* Participants must be aged 18 and above
* Participants who meet the safety criteria for undergoing an MRI scan
* Participants who are able to fit inside the scanner
* Participants must be able to give fully informed consent
* Participants must be mobile enough to be positioned onto the FCI scanner couch

Exclusion Criteria:

* Patients with total hip replacement
* MRI-incompatible conditions, as detected in the MRI safety screening sheet
* Participants under 18 years old
* Participants who are unable to communicate in English
* Participants who are unable to give fully informed consent
* Women who are pregnant
* Restrictions to mobility that would prevent the correct positioning in the scanner
* Participants who suffer from claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Identification of bladder tumours by Field-Cycling Imaging (FCI) scan | At baseline
  Validation of FCI T1 dispersion profiles as a non-invasive technology able to detect bladder tumours.

SECONDARY OUTCOMES:
Differentiation of bladder tumours assessed by Field-Cycling Imaging (FCI) T1 dispersion profiles | At baseline
  Validation of FCI T1 dispersion profiles as a clinical tool for distinguishing non-muscle invasive from muscle-invasive bladder tumours.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Kiltie, Prof, Study Chair — University of Aberdeen

IPD SHARING:
Plan to Share IPD: No